CLINICAL TRIAL: NCT05538507
Title: Efficacy of Chinese Traditional Medicine "Smart Soup" in Cognition and Behavior Regulation in Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Tongji University (Other)
Responsible Party: Principal Investigator, gaojing, Professor, Department of Neurology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Smart Soup
Record Dates: First submitted 2022-04-12; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Alzheimer's disease; Traditional Chinese Medicine; Smart soup
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Medicine, Chinese Traditional; Donepezil; Memantine

STUDY DESIGN:
Intervention Model Description: Patients were divided into 6 groups according to the enrollment criteria, with 30 cases in each group. Group I AD patients were given donepezil 10 mg, memantine 20 mg and smart soup, group II AD patients were given donepezil 10 mg, memantine 20 mg and placebo; group III AD patients were given donepezil 10 mg and smart soup, group IV AD patients were given donepezil 10 mg and and placebo; group V MCI patients were given smart soup, and group VI MCI patients were given placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group I severe AD (Active Comparator): Patients over 40 years of age and eligible for NIA-AA 2011 probable severe AD will be given donepezil 10 mg, memantine 20 mg and smart soup
  Interventions: Drug: smart soup; Drug: Donepezil; Drug: Memantine
- Group II severe AD (Sham Comparator): Patients over 40 years of age and eligible for NIA-AA 2011 probable severe AD will be given donepezil 10 mg, memantine 20 mg and placebo
  Interventions: Drug: Donepezil; Drug: Memantine; Drug: Placebo
- Group III Mild or moderate AD (Active Comparator): Patients over 40 years of age and eligible for NIA-AA 2011 probable mild or moderate AD will be given donepezil 10 mg and smart soup
  Interventions: Drug: smart soup; Drug: Donepezil
- Group IV Mild or moderate AD (Sham Comparator): Patients over 40 years of age and eligible for NIA-AA 2011 probable mild or moderate AD will be given donepezil 10 mg and placebo
  Interventions: Drug: Donepezil; Drug: Placebo
- Group V MCI (Active Comparator): Patients over 40 years of age and eligible for NIA-AA 2011 probable MCI will be given smart soup
  Interventions: Drug: smart soup
- Group VI MCI (Sham Comparator): Patients over 40 years of age and eligible for NIA-AA 2011 probable MCI will be given placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: smart soup — Severe AD, mild or moderate AD and MCI will be given smart soup
  Other Names: traditional chinese medicine
  Arms: Group I severe AD; Group III Mild or moderate AD; Group V MCI
Drug: Donepezil — Severe AD and mild or moderate AD will be given donepezil
  Other Names: donepezil pill
  Arms: Group I severe AD; Group II severe AD; Group III Mild or moderate AD; Group IV Mild or moderate AD
Drug: Memantine — Severe AD will be given memantine
  Other Names: Memantine Pill
  Arms: Group I severe AD; Group II severe AD
Drug: Placebo — patients with MCI will be given placebo
  Arms: Group II severe AD; Group IV Mild or moderate AD; Group VI MCI

SUMMARY:
It is a prospective interventional randomized controlled single center trial. The goal of the trial is to evaluate the efficacy of smart soup on cognition, behavior, biomarkers and safety in Alzheimer's disease (aMCI and dementia).

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia and places a heavy burden on patients, families, society and healthcare. The drugs that have been marketed worldwide for the treatment of AD so far can only delay but not reverse the course of the disease, and the current drug development is all directed at a single target, while the onset of AD is the result of a combination of multiple factors, which is an important reason why so many drugs have faltered. The investigators need to find new multi-target intervention pathways from another perspective.

The advantage of Chinese medicine is multi-target and multi-factor regulation, which has advantages in treating complex diseases. The combination of ancient smart soup with donepezil was able to significantly improve the cognitive function in demented animals. Smart Soup is prepared from three herbs: Rhizoma Acori Tatarinowii, Poria cum Radix Pini, Radix Polygalae. These three herbs are each 15 grams and ground into a very fine powder. This approach reduced the formation of characteristic pathological changes at the pathological level, therefore, the combination of ancient Chinese medicine formulae with modern medical treatment may bring new hope to the treatment of demented patients.

The main design of this study are following: Patients over 40 years of age and eligible for NIA-AA 2011 probable AD and probable MCI were included in this study and were divided into 6 groups of 30 patients each. Group I AD patients were given donepezil 10 mg, memantine 20 mg and smart soup, group II AD patients were given donepezil 10 mg, memantine 20 mg and placebo; group III AD patients were given donepezil 10 mg and smart soup, group IV AD patients were given donepezil 10 mg and placebo; group V mild cognitive impairment (MCI) patients were given smart soup, and group VI MCI patients were given placebo.

Evaluations were set before enrollment, every three months till one year and the evaluators were single-blind. The scales involved in the evaluation of cognitive function and quality of life, sleep condition, and emotional behavior included ADAS-cog, MMSE, CDR, ADL, CMAI, NPI, and EQ-5D, which were evaluated five times. MRI, EEG, blood oxidative stress indicators, and biological markers were collected at the same time at enrollment and at the end of the study. Genotype collection was completed at enrollment. Safety was also evaluated with monthly testing of ECG, routine blood, liver and kidney function, urinary routine, and recording of side effects.

ELIGIBILITY:
Inclusion Criteria:

* NIA-AA 2011 AD probable Alzheimer's disease, mild to moderate, stable use donepezil 10mg/d for 3 months
* NIA-AA 2011 AD probable Alzheimer's disease, severe, stable use donepezil 10mg/d and memantine 20mg/d for 3 months
* NIA-AA 2011 MCI probable criteria
* stable care giver
* Traditional Chinese medicine diagnosis: pixu tanzhuo

Exclusion Criteria:

* Severe systemic disease (heart, liver ,kidney function failure)
* contradictions of MRI examination

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Changes of cognitive screening | Through study completion, an average of 1 years
  Using the neuropsychological scale, mini-mental state examination (MMSE,0-30), to assess every three months after trial entry
Changes of comprehensive cognitive assessment | Through study completion, an average of 1 years
  Use the neuropsychological scales, Alzheimer's Disease Assessment Scale-Cognitive section (ADAS-cog 0-75)， to assess every three months after trial entry
Changes in the degree of dementia | Through study completion, an average of 1 years
  Use the neuropsychological scales, CDR(0-3), to assess every three months after trial entry
Changes in behavior | Through study completion, an average of 1 years
  Use the Cohen-Mansfield Agitation Inventory (CMAI，29-203) to assess every three months after trial entry
Changes in Psychiatric symptoms | Through study completion, an average of 1 years
  Use the Neuropsychiatric Index (NPI) to assess every three months after trial entry
Changes of daily living skills | Through study completion, an average of 1 years
  Use Activity of Daily Living Scale（ADL，20-80）to assess every three months after trial entry
Changes in health status | Through study completion, an average of 1 years
  Use EuroQoL 5-dimension (EQ-5D,0-100) to assess every three months after trial entry
Tau and Beta-amyloid biomarkers in CSF and plasma | Through study completion, an average of 1 years
  Concentration ( pg/mL) of beta-amyloid, tau and phospho-tau in cerebrospinal fluid (CSF) and plasma of patients with dementia and controls
Magnetic resonance imaging and Electroencephalogram（EEG） | Through study completion, an average of 1 years
  Evaluate the imaging and EEG changes of dementia patients. Specifically, EEG can be used to monitor the activity of brain waves in different parts of the cerebral cortex (e.g. power in alpha band, distribution and power of slow theta/delta waves etc.)
Oxidative stress markers in blood | Through study completion, an average of 1 years
  Concentration of Dopamine in blood of patients with dementia and controls
Alterations of neurotransmitters in the blood | Through study completion, an average of 1 years
  Concentration (ng/ml) of 5-hydroxy tryptamine (HT) in blood of patients with dementia and controls

CONTACTS AND LOCATIONS:
Overall Officials: Jing Gao, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hou Y, Wang Y, Zhao J, Li X, Cui J, Ding J, Wang Y, Zeng X, Ling Y, Shen X, Chen S, Huang C, Pei G. Smart Soup, a traditional Chinese medicine formula, ameliorates amyloid pathology and related cognitive deficits. PLoS One. 2014 Nov 11;9(11):e111215. doi: 10.1371/journal.pone.0111215. eCollection 2014. PMID 25386946
- [Background] Wang Y, Wang Y, Sui Y, Yu H, Shen X, Chen S, Pei G, Zhao J, Ding J. The combination of aricept with a traditional Chinese medicine formula, smart soup, may be a novel way to treat Alzheimer's disease. J Alzheimers Dis. 2015;45(4):1185-95. doi: 10.3233/JAD-143183. PMID 25690664
- [Background] Ling Y, Li Z, Chen M, Sun Z, Fan M, Huang C. Analysis of multiple constituents in Cong-Ming-Tang, a Chinese herbal formula for the treatment of amnesia, by high-performance liquid chromatography with quadrupole time-of-flight mass spectrometry. Phytochem Anal. 2013 Nov-Dec;24(6):677-88. doi: 10.1002/pca.2454. Epub 2013 Jul 9. PMID 23839964
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250